CLINICAL TRIAL: NCT03136237
Title: A Phase 1 Study to Evaluate the Effect of BCX7353 on the Single Dose Pharmacokinetics of the P-gp Substrate Digoxin and the BCRP Substrate Rosuvastatin and the Effect of the P-gp Inhibitor Cyclosporine on the Single Dose Pharmacokinetics of BCX7353
Brief Title: A Drug-Drug Interaction Study to Evaluate Drug Transporter Interactions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: BioCryst Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCX7353-105
Record Dates: First submitted 2017-04-24; First posted 2017-05-02 (Actual); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Hereditary Angioedema
MeSH Terms: conditions — Angioedemas, Hereditary | interventions — berotralstat; Digoxin; Rosuvastatin Calcium; Cyclosporine

STUDY DESIGN:
Intervention Model Description: 3 parallel treatment assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Day 1: Digoxin 0.25 mg oral dose Day 11-18: BCX7353 350 mg oral dose Day 19: Digoxin 0.25 mg oral dose and BCX7353 350 mg oral dose Day 20-21: BCX7353 350 mg oral dose
  Interventions: Drug: BCX7353; Drug: Digoxin; Drug: BCX7353 + digoxin
- Cohort 2 (Experimental): Day 1: Rosuvastatin 10 mg oral dose Day 7-14: BCX7353 350 mg oral dose Day 15: Rosuvastatin 10 mg oral dose and BCX7353 350 mg oral dose Day 16: BCX7353 350 mg oral dose
  Interventions: Drug: BCX7353; Drug: Rosuvastatin; Drug: rosuvastatin + BCX7353
- Cohort 3 (Experimental): Day 1: BCX7353 350 mg oral dose Day 14: single oral dose of Cyclosporine 600 mg and BCX7353 350 mg
  Interventions: Drug: BCX7353; Drug: Cyclosporine + BCX7353

INTERVENTIONS:
Drug: BCX7353 — Day 11-18 for Cohort 1, Day 7-14 for Cohort 2, Day 1 for Cohort 3
Drug: Digoxin — Day 1 of Cohort 1
  Arms: Cohort 1
Drug: BCX7353 + digoxin — Day 19 of Cohort 1
  Arms: Cohort 1
Drug: Rosuvastatin — Day 1 of Cohort 2
  Arms: Cohort 2
Drug: rosuvastatin + BCX7353 — Day 15 of Cohort 1
  Arms: Cohort 2
Drug: Cyclosporine + BCX7353 — Day 14 of Cohort 3
  Arms: Cohort 3

SUMMARY:
This is an open-label, three part study to evaluate the effect of BCX7353 on drug transporters as well as the effect of an inhibitor of drug transport on BCX7353.

DETAILED DESCRIPTION:
This is a single center, open-label, fixed-sequence, drug interaction study to evaluate the effect of BCX7353 on the pharmacokinetics of the P-gp substrate digoxin and the BCRP substrate rosuvastatin, as well as the effect of the P-gp inhibitor cyclosporine on the pharmacokinetics of BCX7353.

It is planned that 54 subjects will be enrolled into 3 cohorts of 18 subjects each. Cohort 1 will evaluate the effects of multiple doses of BCX7353 on single-dose pharmacokinetics of digoxin. Cohort 2 will evaluate the effect of multiple doses of BCX7353 on the pharmacokinetics of rosuvastatin. Cohort 3 will evaluate the effect of a single dose of cyclosporine on the pharmacokinetics of BCX7353. Cohorts may be dosed in parallel or in any order.

ELIGIBILITY:
Key Inclusion Criteria:

* written informed consent
* acceptable birth control measures for male subjects and women of childbearing potential
* creatinine clearance of at least 80 mL/min by Cockcroft-Gault equation
* complies with all required study procedures and restrictions

Key Exclusion Criteria:

* clinically significant medical history, current medical or psychiatric condition
* clinically significant ECG finding, vital sign measurement or laboratory/urinalysis abnormality at screening or baseline
* current use, or use of any prescribed or over the counter medication, vitamins or herbal products within 14 days of Day 1
* use of medication that is known to inhibit or induce metabolic enzymes or transporters within 30 days of dosing
* participation in any other investigational drug study within 90 days of screening
* recent or current history of alcohol or drug abuse
* regular recent use of tobacco or nicotine products
* positive serology for HBV, HCV, or HIV
* pregnant or nursing
* donation or loss of greater than 400 mL of blood within the previous 3 months
* history of severe hypersensitivity to any medicinal product
* for subjects enrolled in cohort 1, current use of antibiotics or probiotics, or use within 6 months prior to Day 1

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2017-02-17 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Cmax of probe substrate | plasma pharmacokinetic parameters are based on blood sampling over a 48 - 72 hour period
AUClast of probe substrate | plasma pharmacokinetic parameters are based on blood sampling over a 48 - 72 hour period
AUCinf of probe substrate | plasma pharmacokinetic parameters are based on blood sampling over a 48 - 72 hour period

SECONDARY OUTCOMES:
adverse events | absolute and change from baseline through end of study, approximately 30 days
laboratory analyses | absolute and change from baseline through end of study, approximately 30 days
vital signs | absolute and change from baseline through end of study, approximately 30 days
physical examination findings | absolute and change from baseline through end of study, approximately 30 days
electrocardiograms | absolute and change from baseline throughend of study, approximately 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Firas Almazedi, MBChB, Msc, CPI, Principal Investigator — Covance Clinical
Locations (1):
- Covance CRU, Leeds, United Kingdom